CLINICAL TRIAL: NCT03634956
Title: Reversal of Rocuronium-Induced Neuromuscular Blockade by Sugammadex Increase for Efficiency of Intraoperative Neural Monitoring in the Thyroid Surgery
Brief Title: Effect of IONM on Efficacy and Safety Using Sugammadex in Thyroid Surgery
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Lütfiye Nuri Burat Government Hospital (Other Government)
Responsible Party: Principal Investigator, TURGUT DONMEZ, Principal investigator, Lütfiye Nuri Burat Government Hospital
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: BakirköyEAH 1
Record Dates: First submitted 2018-08-13; First posted 2018-08-17 (Actual); Last update posted 2018-08-20 (Actual); Status verified 2018-08

CONDITIONS: Vocal Cord Paralysis; Recurrent Laryngeal Nerve
Keywords: multinoduler goitre; thyroid cancer; sugammadex sodium; intraoperative nerve monitorization
MeSH Terms: conditions — Vocal Cord Paralysis; Thyroid Neoplasms

STUDY DESIGN:
Intervention Model Description: Group A. Sugammadex sodium-IONM in thyroid surgery Group B.Standart technique-IONM in thyroid surgery
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Group I.IONM in thyroid surgery (Experimental): Group I.IONM in thyroid surgery.Once the vagus has been detected,nerve conduction data will be detected with IONM. If the muscle relaxant effect is not detected, it will be detected with TOF device.
  Interventions: Drug: Group B. Sugammadex sodium-IONM

INTERVENTIONS:
Drug: Group B. Sugammadex sodium-IONM — Group B.the vagal nerve is detected and then 2 mg / kg of sugammadex sodium is administered to remove the muscle relaxant effect
  Other Names: Sugammadex sodium intervention group

SUMMARY:
Thyroidectomy is a frequently performed surgeon by the head and neck and endocrine surgeons. In recent years, surgical techniques and technological developments have resulted in a significant reduction in complication rates. Despite these advances, there is still a great deal of anxiety about the sound problems that can be experienced in patients after surgery. In the past years,the investigators have tried to prevent recurrent nerve paralysis by using intraoperative nerve monitoring (IONM). The use of IONM has begun to be preferred by many surgeons in the investigator's country. However, the use of IONM decreases the number of recurrent nerve paralysis are still being discussed and many studies have been done. In this study, it is aimed to prevent the formation of recurrent nerve paralysis in order to safely carry out the IONM by removing the effects of neuromuscular blockade drugs using sugammadex sodium medicine in the thyroidectomy operations.

DETAILED DESCRIPTION:
Patients who will undergo thyroidectomy using the IONM in the General Surgery Clinic of Istanbul, Bakırköy Dr.Sadi Konuk Training and Research Hospital. In this prospective observational clinical trial, the patients will be divided into two groups and the study will be performed as randomize. Randomization Patients who arrive consecutively, will be included in the study group (Group I IONM, group B IONM-sugammadex sodium). In both groups, anesthesia induction should be done with 3 mg / kg propofol, 2 ugr / kg fentanyl, 0.6 mg / kg rocuronium bromide, as the intubation tube, the number appropriate for the patient, After reaching the throat loom, the patient is entrapped and then the operation is started. After reaching the thyroid loin and hanging the throid with the swab sutures, the lobe is taken out with the finger maneuver and then the vascular nerve packet is dissected and the vagal nerve is exposed. IONM(Medtronic-NIM) were detected in the recurrent nerve thyroglossal groove and 100 microvolts or more were measured with nerve monitoring. + Acceptance of resection was started and IONM After the intubation of the group B-sugammadex sodium was started, the left hand ulnar sinus TOF-Guard device was placed and operation started. After reaching the thyroid loops and hanging the throids with hanging sutures and removing the lobe with finger maneuver, the vascular nerve was disassembled and the vagal nerve was dislocated. Then the electrical value was recorded with IONM and sugammadex sodium 2 mg / kg was made. and the TOF response at 4th minute is over 90% of the value to be measured and if the IONM is 100 microvolts higher, the recurrent nerve is found in the troglossal groove and the nerve is followed with the IONM and the resection procedure is started and the tirodidectomy will be performed. V0: vagal nerve initial value; V1: value before troid resection; V2: value after troid resection; R1: value after troid resection, R2: value after troid resection. Preoperative and postoperative vocal cord examination will be examined by otolaryngologist. Size, weight, sex, ASA scores, operation times, complications will be recorded. If there is no signal in RLN with intraoperative IONM and RLN paralysis will be accepted if there is inactivity in the vocal cord at the 1st postoperative ENT specialist vocal cord examinations. RLN paralysis will be accepted if there is inactivity in the cord at the vocal cord examination of the postoperative specialist ENT specialist. The ENT specialist and general surgeon will follow up and if the vocal cord is still in motion, the permanent RLN will be considered a paralysis.

ELIGIBILITY:
Inclusion Criteria:

* Clinical diagnosis of Multinodular goiter,
* Clinical diagnosis of thyroid cancer
* Clinical diagnosis of noduler goatr,
* Clinical diagnosis of basedow Graves disease,

Exclusion Criteria:

* Patients with bleeding diathesis,
* Patients who have previously undergone laryngeal surgery (vocal polyps, nodules or laryngeal cancer),

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 2 (Estimated)
Dates: Start 2018-08-14 (Actual); Primary Completion 2019-02-14 (Estimated); Study Completion 2019-03-14 (Estimated)

PRIMARY OUTCOMES:
Vocal cord paralysis | postop 15th days
  postoperative vocal cord examination will be performed and the recurrent laryngeal nerve will be examined.

SECONDARY OUTCOMES:
vagal nerve conduction value(V1) | 15 to 45 minutes of surgery
  V1: value to receive enough nerve conduction for IONM use from the vagus nerve
vagal nerve conduction value after lob resection(V2) | 30 to 90 minutes of surgery
  V2:Vagus value after resection of thyroid lobe
first detected vagal nerve conduction value(V0) | 5 to 25 minutes of surgery
  initial value after vagus sinus is detected
TOF time | 10 to 90 minutes of surgery
  the time that the muscle relaxant is shown by the peripheral nerve stimulator whose effect has disappeared.TOF>0.9

CONTACTS AND LOCATIONS:
Overall Officials: Turgut Donmez, surgeon, Principal Investigator — Lütfiye Nuri Burat Goverment Hastanesi
Locations (1):
- Lutfiye NBGH, Istanbul, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: Yes
Patients who are accepted to participate in the study will be gathered in the pool. The patients' data will be entered on the computer. The computer and patients will be randomized and set up on the day of surgery. The preop, perop and postop data of the patients will be recorded on the computer.
Supporting Information: Study Protocol, SAP, ICF, CSR, Analytic Code
Time Frame: 14.08.2018-14.02.2019
Access Criteria: the study data will be stored securely on the researcher's turgut donmez personal computer. It will be available to researchers participating in the study alone

REFERENCES:
- [Background] Empis de Vendin O, Schmartz D, Brunaud L, Fuchs-Buder T. Recurrent Laryngeal Nerve Monitoring and Rocuronium: A Selective Sugammadex Reversal Protocol. World J Surg. 2017 Sep;41(9):2298-2303. doi: 10.1007/s00268-017-4004-9. PMID 28349321
- [Background] Barczynski M, Konturek A, Cichon S. Randomized clinical trial of visualization versus neuromonitoring of recurrent laryngeal nerves during thyroidectomy. Br J Surg. 2009 Mar;96(3):240-6. doi: 10.1002/bjs.6417. PMID 19177420